CLINICAL TRIAL: NCT01778738
Title: Glycaemia, Insulin Secretion and Action in Morbidly Obese Subjects With Type 2 Diabetes After Sleeve Gastrectomy and Roux-en-Y Gastric Bypass: A Randomised Single Centre Study
Brief Title: Type 2 Diabetes After Sleeve Gastrectomy and Roux-en-Y Gastric Bypass: A Randomised Single Centre Study
Acronym: OSEBERG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset i Vestfold HF (Other)
Responsible Party: Principal Investigator, Dag Hofsø, Prinsipal Investigator, Sykehuset i Vestfold HF
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012/1427b
Record Dates: First submitted 2012-12-03; First posted 2013-01-29 (Estimated); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Type 2 Diabetes; Morbid Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity, Morbid | interventions — Bariatric Surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sleeve gastrectomy (Experimental): Sleeve gastrectomy.
  Interventions: Procedure: Bariatric surgery, either gastric bypass surgery or sleeve gastrectomy; Procedure: Sleeve gastrecomy
- Gastric bypass (Experimental): Gastric bypass surgery.
  Interventions: Procedure: Bariatric surgery, either gastric bypass surgery or sleeve gastrectomy; Procedure: Bastric bypass
- Control group (No Intervention): This is an extra control group without diabetes. All subjects are morbidly obese patients recruited from the Morbid Obesity Centre.

INTERVENTIONS:
Procedure: Bariatric surgery, either gastric bypass surgery or sleeve gastrectomy — Vertical sleeve gastrectomy or a gastric bypass surgery in morbidly obese individuals with type 2 diabetes. Random allocation to surgical intervention
  Arms: Gastric bypass; Sleeve gastrectomy
Procedure: Sleeve gastrecomy — Vertical sleeve gastrectomy
  Arms: Sleeve gastrectomy
Procedure: Bastric bypass — Gastric bypass surgery
  Arms: Gastric bypass

SUMMARY:
Glycaemia, insulin secretion and action in morbidly obes subjects with type 2 diabetes after sleeve gastrectomy ond Roux-en-Y gastric bypass: A randomised single centre study.

DETAILED DESCRIPTION:
The Roux-en-Y gastric bypass operation combines restrictive and malabsorptive principles. It is the most commonly performed bariatric procedure worldwide (~ 50 %). Vertical (sleeve) gastrectomy on the other hand, is a purely restrictive procedure and has gained popularity and is now accepted as a valid procedure accounting for approximately five percent of the bariatric procedures performed worldwide.

The remission rate of type 2 diabetes one to two years after bariatric surgery is approximately 70%. Some studies have indicate that the remission rate of type 2 diabetes is higher after gastric bypass than after sleeve gastrectomy. Other studies indicate a similar effect on the reduction in HbA1c.

Weight reduction is comparable between gastric bypass and sleeve gastrectomy although some evidence suggets a larger weight loss following gastric bypass surgery. Larger weight loss can clearly contribute to somewhat greater improvement in glucose homeostasis after gastric bypass than after sleeve gastrectomy. Still, one might speculate that changes in gut hormones may contribute to higher remission rates of type 2 diabetes after gastric bypass than after sleeve gastrectomy.

Improved β-cell function observed after gastric bypass surgery may be linked to higher postprandial levels of Glucagonlike peptide 1 as seen after gastric bypass surgery. Beta cell function has, to our knowledge, only been addressed in one previous study after sleeve gastrectomy, with the authors reporting an increased first-phase insulin secretion three days after the procedure. Although several studies have addressed changes in gastrointestinal hormones the incretin effect on insulin secretion after gastric bypass has been estimated in only a few studies. To the best of our knowledge the incretin effect on insulin secretion after sleeve gastrectomy remains unexplored.We are aware of four ongoing randomised controlled trials comparing the effect of gastric bypass and sleeve gastrectomy on several endpoints including weight and comorbidities (ClinicalTrial.gov identifiers: NCT00722995, NCT00356213, NCT00793143, and NCT00667706). However, these studies include both subjects with and with-out type 2 diabetes and are therefore not powered to detect between-group differences in HbA1c and beta-cell function in the diabetic patients.

In conclusion, the effect of gastric bypass and sleeve gastrectomy on glycaemia is not fully elucidated. Moreover, the impact of altered beta-cell function post surgery needs to be explored. We hypothesise that greater improvement in beta-cell function after gastric bypass than after sleeve gastrectomy translates into better glycaemic control in subjects with type 2 diabetes one year after surgery.

ELIGIBILITY:
Inclusion criteria

* Previously verified BMI ≥35.0 kg/m2 and current BMI ≥33.0 kg/m2
* HbA1c ≥6.5 % or use of anti-diabetic medications with HbA1c ≥6.1 %
* Age ≥18 years

Exclusion criteria

* Not able to give informed consent
* Previously major abdominal surgery (appendectomy, laparoscopic cholecystectomy or gynaecological procedures not included)
* Severe endocrine-, heart-, lung-, liver- and kidney disease, cancer and other medical conditions associated with significantly increased risk of peri- and postoperative complications
* Drug or alcohol addiction
* Reduced compliance due to severe mental and psychiatric conditions
* Pregnancy
* Serum autoantibodies against glutamic acid decarboxylase (GAD) or tyrosine phosphatase (IA2)
* Regular use (a total of 3 months cumulative use in the last 12 months) or treatment the past two months with systemic corticosteroids
* Severe gastroesophageal reflux disease defined as Los Angeles classification grade > B, Barrett's oesophagus and/or hiatus hernia >5 cm
* Elevated esophageal pressure (DCI >5000 mmHg*sec*cm) and symptoms of dysphagia and/or painful swallowing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2022-11 (Actual)

PRIMARY OUTCOMES:
Remission of type 2 diabetes. | One year
  HbA1c below or equal to 6.0 % in the absence of glucose lowering drug therapy
Beta-cell function | One Year
  Disposition index calculated using glucose and insulin data obtained from a frequently sampled intravenous glucose tolerance test.

SECONDARY OUTCOMES:
Glycaemic control | Five weeks to five years
  HbA1c
Insulin secretion | Five weeks to five years
  Fasting and stimulated levels of glucose, insulin, C-peptide and proinsulin after an oral glucose load will be used for the calculation of insulin secretion.
Insulin sensitivity | Five weeks to five years
  Fasting and stimulated levels of glucose, insulin and C-peptide after an oral glucose load will be used for the calculation of insulin sensitivity.
Anti-diabetic medication | Five weeks to five years
  Use of glucose lowering agents
Body weight | Five weeks to five years
  Body weight (kg and kg/m2)
Body composition | Five weeks to five years
  Measured by DEXA and bioelectrical impedance analysis
Blood pressure | Five weeks to five years
  Resting and 24-h ambulatory systolic and diastolic blood pressure
Pulse wave velocity | Five weeks to five years
  The Sphygmocor system (Artcor, Sidney, Australia) and a single high-fidelity applanation tonometer (Millar®) will be used to measure pulse wave velocity.
Lipidemia | Five weeks to five years
  Cholesterol and triglyceride levels
Obstructive sleep apnoea | Five weeks to five years
  The ApneaLink Plus was used for the calculation of apnoeas and hypopnoeas during sleep.
Proteinuria | Five weeks to five years
  Urine protein-to-creatinine and albumin-to-creatinine ratios
Gastroesophageal reflux disease | One to five years
  Gastroesophageal reflux disease will be diagnosed using upper endoscopy, 24 hour intra-oesophageal pH monitoring and symptom scores.
Gastroesophageal motility disorders | One to five years
  High-resolution manometry
Fatty liver disease | One to five years
  MRI (Siemens Aera 1.5 T) and Chemical Shift Imaging18 will be used to quantify the fat-fraction content of the liver.
Gut microbiota | One to five years
  Microbial composition and diversity and quantification of organic acids and DNA extraction and metagenome data analysis.
Physical activity | Five weeks to five years
  Measured and self-reported physical activity
Energy intake and eating behaviour | Five weeks to five years
  Food frequency questionnaire, food tolerance questionnaire, power of food scale and binge eating scale
Health related quality of life | Five weeks to five years
  Short Form Quality of Life questionnaire (SF-36) v. 2.0
Obesity-related symptoms | Five weeks to five years
  Impact on Weight Questionnaire IWQOL-Lite and Weight-Related Symptom Measure (WRSM)
Psychological distress | Five weeks to five years
  Beck Depression Inventory
Bone mineral density | Five weeks to five years
  DEXA scan
Dumping syndrome | Five weeks to five years
  Arts' questionnaire
Vitamin and mineral deficiencies | Five weeks to five years
  Vitamin (B1, B9, B12, D) and mineral (calcium, iron) levels in blood.

CONTACTS AND LOCATIONS:
Overall Officials: Jøran Hjelmesæth, Professor, Study Chair — Head of the Morbid Obesity Centre
Locations (1):
- The Morbid Obesity Center, Vestfold Hospital Trust, Tønsberg, Vestfold, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hofso D, Fatima F, Borgeraas H, Birkeland KI, Gulseth HL, Hertel JK, Johnson LK, Lindberg M, Nordstrand N, Cvancarova Smastuen M, Stefanovski D, Svanevik M, Gretland Valderhaug T, Sandbu R, Hjelmesaeth J. Gastric bypass versus sleeve gastrectomy in patients with type 2 diabetes (Oseberg): a single-centre, triple-blind, randomised controlled trial. Lancet Diabetes Endocrinol. 2019 Dec;7(12):912-924. doi: 10.1016/S2213-8587(19)30344-4. Epub 2019 Oct 31. PMID 31678062
- [Result] Borgeraas H, Hjelmesaeth J, Birkeland KI, Fatima F, Grimnes JO, Gulseth HL, Halvorsen E, Hertel JK, Hillestad TOW, Johnson LK, Karlsen TI, Kolotkin RL, Kvan NP, Lindberg M, Lorentzen J, Nordstrand N, Sandbu R, Seeberg KA, Seip B, Svanevik M, Valderhaug TG, Hofso D. Single-centre, triple-blinded, randomised, 1-year, parallel-group, superiority study to compare the effects of Roux-en-Y gastric bypass and sleeve gastrectomy on remission of type 2 diabetes and beta-cell function in subjects with morbid obesity: a protocol for the Obesity surgery in Tonsberg (Oseberg) study. BMJ Open. 2019 Jun 4;9(6):e024573. doi: 10.1136/bmjopen-2018-024573. PMID 31167860
- [Result] Lorentzen J, Medhus AW, Hertel JK, Borgeraas H, Karlsen TI, Kolotkin RL, Sandbu R, Sifrim D, Svanevik M, Hofso D, Seip B, Hjelmesaeth J. Erosive Esophagitis and Symptoms of Gastroesophageal Reflux Disease in Patients with Morbid Obesity with and without Type 2 Diabetes: a Cross-sectional Study. Obes Surg. 2020 Jul;30(7):2667-2675. doi: 10.1007/s11695-020-04545-w. PMID 32193740
- [Result] Hofso D, Hillestad TOW, Halvorsen E, Fatima F, Johnson LK, Lindberg M, Svanevik M, Sandbu R, Hjelmesaeth J. Bone Mineral Density and Turnover After Sleeve Gastrectomy and Gastric Bypass: A Randomized Controlled Trial (Oseberg). J Clin Endocrinol Metab. 2021 Jan 23;106(2):501-511. doi: 10.1210/clinem/dgaa808. PMID 33150385
- [Result] Fatima F, Hjelmesaeth J, Hertel JK, Svanevik M, Sandbu R, Smastuen MC, Hofso D. Validation of Ad-DiaRem and ABCD Diabetes Remission Prediction Scores at 1-Year After Roux-en-Y Gastric Bypass and Sleeve Gastrectomy in the Randomized Controlled Oseberg Trial. Obes Surg. 2022 Mar;32(3):801-809. doi: 10.1007/s11695-021-05856-2. Epub 2022 Jan 4. PMID 34982397
- [Result] Fatima F, Hjelmesaeth J, Birkeland KI, Gulseth HL, Hertel JK, Svanevik M, Sandbu R, Smastuen MC, Hartmann B, Holst JJ, Hofso D. Gastrointestinal Hormones and beta-Cell Function After Gastric Bypass and Sleeve Gastrectomy: A Randomized Controlled Trial (Oseberg). J Clin Endocrinol Metab. 2022 Jan 18;107(2):e756-e766. doi: 10.1210/clinem/dgab643. PMID 34463768
- [Result] Seeberg KA, Borgeraas H, Hofso D, Smastuen MC, Kvan NP, Grimnes JO, Lindberg M, Fatima F, Seeberg LT, Sandbu R, Hjelmesaeth J, Hertel JK. Gastric Bypass Versus Sleeve Gastrectomy in Type 2 Diabetes: Effects on Hepatic Steatosis and Fibrosis : A Randomized Controlled Trial. Ann Intern Med. 2022 Jan;175(1):74-83. doi: 10.7326/M21-1962. Epub 2021 Nov 30. PMID 34843380
- [Result] Lorentzen J, Medhus AW, Hofso D, Svanevik M, Seip B, Hjelmesaeth J. Sleeve Gastrectomy Confers Higher Risk of Gastroesophageal Reflux Disease Than Gastric Bypass: A Randomized Controlled Trial From the Oseberg Reflux Working Group. Gastroenterology. 2021 Dec;161(6):2044-2046.e4. doi: 10.1053/j.gastro.2021.08.021. Epub 2021 Aug 20. No abstract available. PMID 34419459
- [Derived] Wagen Hauge J, Borgeraas H, Birkeland KI, Johnson LK, Hertel JK, Hagen M, Gulseth HL, Lindberg M, Lorentzen J, Seip B, Kolotkin RL, Svanevik M, Valderhaug TG, Sandbu R, Hjelmesaeth J, Hofso D. Effect of gastric bypass versus sleeve gastrectomy on the remission of type 2 diabetes, weight loss, and cardiovascular risk factors at 5 years (Oseberg): secondary outcomes of a single-centre, triple-blind, randomised controlled trial. Lancet Diabetes Endocrinol. 2025 May;13(5):397-409. doi: 10.1016/S2213-8587(24)00396-6. Epub 2025 Apr 1. PMID 40185112
- [Derived] Svanevik M, Lorentzen J, Borgeraas H, Sandbu R, Seip B, Medhus AW, Hertel JK, Kolotkin RL, Smastuen MC, Hofso D, Hjelmesaeth J. Patient-reported outcomes, weight loss, and remission of type 2 diabetes 3 years after gastric bypass and sleeve gastrectomy (Oseberg); a single-centre, randomised controlled trial. Lancet Diabetes Endocrinol. 2023 Aug;11(8):555-566. doi: 10.1016/S2213-8587(23)00127-4. Epub 2023 Jul 3. PMID 37414071
- [Derived] Barstad LH, Johnson LK, Borgeraas H, Hofso D, Svanevik M, Smastuen MC, Hertel JK, Hjelmesaeth J. Changes in dietary intake, food tolerance, hedonic hunger, binge eating problems, and gastrointestinal symptoms after sleeve gastrectomy compared with after gastric bypass; 1-year results from the Oseberg study-a randomized controlled trial. Am J Clin Nutr. 2023 Mar;117(3):586-598. doi: 10.1016/j.ajcnut.2022.11.016. Epub 2022 Dec 22. PMID 36811476
- [Derived] Seeberg KA, Hofso D, Borgeraas H, Grimnes JO, Fatima F, Seeberg LT, Kvan NP, Svanevik M, Hertel JK, Hjelmesaeth J. Association between hepatic steatosis and fibrosis with measures of insulin sensitivity in patients with severe obesity and type 2 diabetes - a cross-sectional study. BMC Gastroenterol. 2022 Nov 7;22(1):448. doi: 10.1186/s12876-022-02550-0. PMID 36336684